CLINICAL TRIAL: NCT06378541
Title: Virtual Hope Box Enhanced Facilitation in High-Risk Suicidal Veterans
Brief Title: Smartphone App Enhanced Facilitation Among Veterans in a Mental Health Inpatient Setting (Project HOPE)
Acronym: Project HOPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SDR 21-267
Record Dates: First submitted 2024-04-15; First posted 2024-04-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Suicide Prevention; Suicide Attempt; Suicide Ideation
Keywords: smartphone application; suicide prevention; virtual hope box; veterans
MeSH Terms: conditions — Suicide Prevention; Suicide, Attempted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Hope Box Enhanced Facilitation (VHB-EF) (Experimental): The VHB-EF intervention has two phases: (1) The in-person inpatient phase involves a single, one-on-one, 60-minute session delivered by the study interventionist prior to hospital discharge. During this session, the interventionist will obtain access to the participant's personal phone and assist them in downloading the VHB app. The interventionist will provide education about the app and personalized behavioral practice for each component of the app. They will also address strategies to enhance app use. In addition, participants will review a list of Veteran mental health resources, community services, Veteran service organizations, and other Veteran social support services available to Veterans in the area. (2) The remote-delivery phase builds on the work begun in the hospital via 2 follow-up phone contacts within 14 days following discharge, during which the study interventionist will monitor risk, review/revise VHB content, and support app use and outpatient treatment engagement.
  Interventions: Behavioral: Virtual Hope Box Enhanced Facilitation
- Enhanced Usual Care (EUC) (Active Comparator): The EUC condition will involve a one-on-one, 30-minute session delivered by the study interventionist prior to hospital discharge, during which the interventionist will review Veteran mental health resources, community services, Veteran service organizations, and other Veteran social support services available to Veterans in the area. The EUC session will remain focused only on reviewing the standardized list of Veteran and community services; no counseling will be provided, and the list provided by the study interventionist does not include non-services (i.e., does not list any smartphone applications, including the VHB app).
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Virtual Hope Box Enhanced Facilitation — The VHB-EF intervention has two phases: (1) The in-person inpatient phase involves a single, one-on-one, 60-minute session delivered by the study interventionist prior to hospital discharge. During this session, the interventionist will obtain access to the participant's personal phone and assist them in downloading the VHB app. The interventionist will provide education about the app and personalized behavioral practice for each component of the app. They will also address strategies to enhance app use. In addition, participants will receive a list of Veteran mental health resources, community services, Veteran service organizations, and other Veteran social support services available to Veterans in the area. (2) The remote-delivery phase builds on the work begun in the hospital via 2 follow-up phone contacts within 14 days following discharge, during which the study interventionist will monitor risk, review/revise VHB content, and support app use and outpatient treatment engagement.
  Other Names: VHB-EF
  Arms: Virtual Hope Box Enhanced Facilitation (VHB-EF)
Behavioral: Enhanced Usual Care — The EUC condition will involve a one-on-one, 30-minute session delivered prior to hospital discharge, during which the study interventionist will review a list of Veteran mental health resources, community services, Veteran service organizations, and other Veteran social support services available to Veterans in the area. The EUC session will remain focused only on reviewing the standardized list of Veteran and community services; no counseling will be provided, and the list provided by the study interventionist does not include non-services (i.e., does not list any smartphone applications, including the VHB app).
  Other Names: EUC
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
This study will test whether a novel intervention, Virtual Hope Box Enhanced Facilitation (VHB-EF), reduces suicide risk in Veterans after discharge from inpatient psychiatric hospitalization. Additionally, this study will also conduct interviews with Veterans and healthcare providers to explore barriers and facilitators to future adoption of the VHB-EF intervention in healthcare settings.

DETAILED DESCRIPTION:
The specific aims of this study are:

Aim 1: To evaluate the effects of VHB-EF for reducing suicide behaviors (primary outcome).

H1: Suicidal Veterans in the VHB-EF arm will be less likely to have suicide behaviors over the 6 months following enrollment compared to those in the EUC condition. The investigators will also examine the effects of VHB-EF on severity of suicidal ideation (secondary outcome).

Aim 2: Examine intervention mechanisms by measuring the effects of VHB-EF on potential mediators, 1) reasons for living, and 2) self-efficacy to (a) cope and (b) refrain from suicide attempts.

H2: VHB-EF Veterans will report higher levels of reasons for living and self-efficacy, compared to EUC. Exploratory sub-aim: The investigators will test the hypothesis that higher levels of reasons for living and self-efficacy will partially mediate the effect of VHB-EF on suicide behaviors over 6-months. Furthermore, the investigators will measure the effects of VHB-EF (vs. EUC) on depressive symptoms and healthcare utilization, and their potential role as mediators of outcomes.

Aim 3: To examine the determinants (barriers and facilitators) of VHB-EF adoption to inform future implementation and sustainability of VHB-EF across the VA. The investigators will conduct qualitative interviews with providers and Veterans to determine the feasibility and acceptability of VHB-EF. This will be used to refine the intervention to maximize the impact of future implementation.

Methods: This is a 2-site randomized effectiveness-implementation hybrid type I trial that will recruit Veterans (N=928) hospitalized for suicidal crises, test this intervention, and gather data to support future implementation. Outcomes will be assessed at 6 weeks, 3 months, and 6 months post-baseline. The study will also include qualitative interviews with providers and Veterans to assess the feasibility and acceptability of VHB-EF.

Significance: This innovative study is the first to test the VHB's impact on suicidal behavior in Veterans during high-risk periods following acute care, addressing a key gap in suicide prevention for this vulnerable group.

ELIGIBILITY:
Inclusion Criteria:

Those enrolled in the RCT component of this study must be:

* 1) Veterans aged 18 or older
* 2) admitted to the inpatient psychiatric unit for a recent suicidal crisis
* 3) medically stable (the patient's medical and psychological fitness [including aggression] to provide informed consent will be determined by a member of the patient's treatment team)
* 4) A score of 3 or greater on the Callahan 6-item cognitive screening.
* 5) report current suicidal ideation (Scale for Suicidal Ideation [SSI]; sum of items 4 and 5 > 0, referencing the week prior to their hospitalization) as reported during the screening interview
* 6) no reported use of the VHB within the past 12-months
* 7) access to a smartphone to download the VHB app

Exclusion Criteria:

Veterans will be found ineligible for the program if:

* 1) do not understand English
* 2) are prisoners
* 3) are unable to provide informed consent
* 4) have profound psychotic symptoms and/or cognitive deficits that would prevent patients from understanding the content of the intervention and/or assessments
* 5) to not have access to a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 928 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
6 month Suicide Behaviors (measured by the Columbia Suicide Severity Rating Scale [C-SSRS]) | 6 months
  Suicide behaviors will be measured by the C-SSRS and will be administered as a semi-structured interview. The definition of suicide behaviors for the primary outcome will consist of any actual suicide attempt or interrupted suicide attempt or aborted suicide attempt during the specified time period.

SECONDARY OUTCOMES:
6 month Suicidal ideation (measured by the Scale for Suicidal Ideation [SSI]-Worst Point) | 6 months
  Worst-point severity of suicidal ideation will be measured by the Scale for Suicidal Ideation (SSI) interview. The total score (sum of the first 19 items) will be used. Scores range from 0 to 38. Increasing scores reflect greater suicide risk.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney L Bagge, PhD MA, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerner JL, Tucker RP, Moscardini EH, Bagge CL, Reger MA. The Virtual Hope Box mobile application: A systematic review of the literature. Suicide Life Threat Behav. 2024 Jun;54(3):501-514. doi: 10.1111/sltb.13061. Epub 2024 Feb 21. PMID 38380558